CLINICAL TRIAL: NCT03189420
Title: Glioma Microenvironment an Exploratory Study
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Raquel Chacon Ruiz Martinez, Principal investigator, PhD, Hospital Sirio-Libanes
Other Study IDs: CAAE 58310716.6.0000.5461
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Glioma of Brain
Keywords: glioma; glioblastoma; low grade tumor
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Transurethral Resection of Bladder; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glioblastoma: Samples of brain tumor diagnosed as glioblastoma
  Interventions: Procedure: Tumor resection
- Low grade glioma: Samples of brain tumor diagnosed as low grade glioma
  Interventions: Procedure: Tumor resection

INTERVENTIONS:
Procedure: Tumor resection — The tumors will be resected in routine therapeutic surgeries
  Other Names: surgery

SUMMARY:
Diffuse glioms are primary brain tumors characterized by infiltrative growth and high heterogeneity, which render the disease mostly incurable. Advances in genetic analysis revealed that molecular and epigenetic alterations predict patients´s overall survival and clinical outcome. However, glioma tumorigenicity is not exclusively caused by its genetic alterations. The crosstalk between tumor cells and the surrounding microenvironment plays a crucial role in modulating glioma growth and aggressiveness. In this sense, to understand the tumor microenvironment would elucidate potential treatment alternatives. The focus will be to evaluate myeloid cells and cytokines levels.

DETAILED DESCRIPTION:
The proposal is to study gene expression and early epigenetic changes in myeloid cells from brain tumors and co-culture experiments. Tough RNA-seq, ATAC-seg and subsequent analysis to monitor the differential gene expression through different time points followed by stimuli. The study will compare the obtained results with sequencing data from microglia of full-fledged human tumor samples (glioblastoma and low grade gliomas). Additionally it will evaluated the immunologic characteristic of the tumor through cytokines levels analysis (TNF-α, IL-4, IL-6, IL-8, IL-10, IL-13, IFN-γ, TGF-β e IL-1ra).

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old with brain tumor
* Patients that will be submitted to brain tumor ressection

Exclusion Criteria:

* Chronic neurodegenerative and inflamatory diseases

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18-65 years old diagnosed with glioblastoma or low grade glioma
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
gene expression changes | 2 years
  Though RNA-seq, ATAC-seg and subsequent analysis we will be able to monitor the differential gene expression through different time points followed by stimuli.

SECONDARY OUTCOMES:
cytokines expression | 2 years
  will evaluate the immunologic characteristic of the tumor through cytokines levels analysis (TNF-α, IL-4, IL-6, IL-8, IL-10, IL-13, IFN-γ, TGF-β e IL-1ra).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sirio Libanes, São Paulo, Sao, Brazil

REFERENCES:
- [Background] Komori T. The 2016 WHO Classification of Tumours of the Central Nervous System: The Major Points of Revision. Neurol Med Chir (Tokyo). 2017 Jul 15;57(7):301-311. doi: 10.2176/nmc.ra.2017-0010. Epub 2017 Jun 8. PMID 28592714
- [Background] Galatro TF, Vainchtein ID, Brouwer N, Boddeke EWGM, Eggen BJL. Isolation of Microglia and Immune Infiltrates from Mouse and Primate Central Nervous System. Methods Mol Biol. 2017;1559:333-342. doi: 10.1007/978-1-4939-6786-5_23. PMID 28063055
- [Background] Quail DF, Joyce JA. The Microenvironmental Landscape of Brain Tumors. Cancer Cell. 2017 Mar 13;31(3):326-341. doi: 10.1016/j.ccell.2017.02.009. PMID 28292436
- [Background] Chiorean R, Berindan-Neagoe I, Braicu C, Florian IS, Leucuta D, Crisan D, Cernea V. Quantitative expression of serum biomarkers involved in angiogenesis and inflammation, in patients with glioblastoma multiforme: correlations with clinical data. Cancer Biomark. 2014;14(2-3):185-94. doi: 10.3233/CBM-130310. PMID 24878820